CLINICAL TRIAL: NCT03116295
Title: A Comparative, Randomized, Open-label, Fasted, Single-dose, 2-way Crossover Bioavailability and Bioequivalence Study of Two Different Sources of Opicapone in Healthy Subjects
Brief Title: Bioavailability and Bioequivalence Study of Two Different Sources of Opicapone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-129
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - 25 mg OPC (Experimental): In Group 1, subjects will receive randomly in Period 1 and 2, either a single 25 mg dose of OPC [AF] or a single 25 mg dose of OPC [NF]. Treatments will be administered in the fasting state, the subjects having fasted for at least 10 hours
  Interventions: Drug: Opicapone (OPC)
- Group 2 - 50 mg OPC (Experimental): In Group 2, subjects will receive randomly on Period 1 and 2, either a single 50 mg dose of OPC [AF], or a single 50 mg dose of OPC [NF]. Treatments will be administered in the fasting state, the subjects having fasted for at least 10 hours
  Interventions: Drug: Opicapone (OPC)

INTERVENTIONS:
Drug: Opicapone (OPC) — Test treatment: 25 mg or 50 mg of OPC hard capsule (new API source NF) Reference treatment: Ongentys® 25 mg or 50 mg of OPC hard capsule (current API source - AF).
  Other Names: Ongentys; BIA 9-1067

SUMMARY:
The purpose of this study is to evaluate the bioavailability and the bioequivalence between two active pharmaceutical ingredient (API) sources of opicapone (OPC) at two different dosage strengths (25 mg and 50 mg) after a single oral dose administration under fasting conditions in healthy male and female subjects.

DETAILED DESCRIPTION:
Single-center, fasted, open-label, randomized, gender-balanced, single-dose, laboratory blinded, two-periods, two-sequence, crossover study in 2 groups of subjects.

In Group 1, subjects will receive randomly in Period 1 and 2, either a single 25 mg dose of OPC approved formulation [AF] or a single 25 mg dose of OPC formulation to be submitted for approval [NF].

In Group 2, subjects will receive randomly on Period 1 and 2, either a single 50 mg dose of OPC (AF), or a single 50 mg dose of OPC (NF

ELIGIBILITY:
Inclusion Criteria:

* Subjects signed and dated the ICF before any study-specific screening procedure.
* Male and female subjects, between 18 and 55 years of age (inclusive).
* BMI between 18 and 30 kg/m² inclusive.
* Subjects have a supine blood pressure (after at least 5 minutes rest in supine position) of: systolic blood pressure ≥90 and <140 mmHg, diastolic blood pressure ≥50 and <90 mmHg and a pulse rate ≥50 and ≤90 bpm (beats per minute).
* Subjects have no clinically relevant abnormal ECG parameters: heart rate ≥50 and ≤90 bpm, PR interval ≤ 220 milliseconds (ms), QRS duration ≤120 ms, QTcB interval ≤450 ms. No clinically relevant pathological findings in the 12-lead ECG.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibodies (HCVab) and anti-HIV antibodies (HIV-1 and HIV-2 Ab) at screening.
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Non-smokers or ex-smokers for at least 3 months.
* If female, the pregnancy test at screening and at admission to each treatment period must be negative.
* Female subjects are of non-childbearing potential (postmenopausal [no menses for at least 1 year] or surgically sterile [tubal ligation, hysterectomy or bilateral oophorectomy]). Female subjects of childbearing potential must use an acceptable method of non-hormonal method of contraception and should be informed of the potential risks associated with becoming pregnant while enrolled within a clinical investigation. Acceptable methods for this study are: intrauterine device, condom or occlusive cap (diaphragm or cervical or vault caps) with spermicide, true abstinence or vasectomized male partner, provided that he is the sole partner of that subject).
* Able to participate, and willing to give written ICF and comply with the study restrictions.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders, or have a clinically relevant surgical history.
* Subjects with clinically relevant neurologic or psychiatric illness.
* Subjects with a history of symptomatic orthostatic hypotension.
* Subjects with clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing) as judged by the Principal investigator.
* Subjects with hereditary galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Subjects with clinically significant findings in laboratory tests, particularly any abnormality in the coagulation tests, or any abnormality in the kidney function tests especially creatinine above 1.2 x upper limit of normal (ULN) and/or liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST],) above 1.25 x ULN confirmed by two repeated measurements, when it is checked during the screening laboratory tests.
* Subjects with a history of relevant atopy or drug hypersensitivity.
* Subjects with a history of alcoholism and/or drug abuse.
* Consumption of more than 14 units of alcohol per week [1 unit of alcohol = 280 ml beer (3-4°) = 100 ml wine (10-12°) = 30 ml spirits (40°)].
* Subjects with a significant infection or known inflammatory process at screening or admission to each treatment period.
* Subjects with acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of screening or admission to each treatment period.
* Use of medicines within 2 weeks prior to the planned first drug administration that may affect the safety or other study assessments, in the investigator's opinion (excluding single use of up to 1000 mg paracetamol).
* Use of any investigational drug or participation in any clinical trial within 30 days or 10 half-life, whatever is longer, prior to the planned first drug administration.
* Donation or receipt of any blood or blood products within the 2 months prior to the planned first drug administration.
* Subjects who are vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Subjects who are unwilling or unable to give written informed consent.
* If female: She is pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration. (Cmax) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Time of the maximum drug concentration (tmax) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Area under the plasma concentration-time curve calculated from time zero (time of drug administration) to the latest time point with a quantifiable plasma concentration (AUC0-t) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent terminal elimination rate constant - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent terminal elimination half-life (t1/2) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent total body clearance (CL/F) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent volume of distribution (V/F) - Period 1 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Maximum observed drug concentration (Cmax) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Time of the maximum drug concentration (tmax) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Area under the plasma concentration-time curve calculated from time zero (time of drug administration) to the latest time point with a quantifiable plasma concentration (AUC0-t) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent terminal elimination rate constant - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent terminal elimination half-life (t1/2) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent total body clearance (CL/F) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables
Apparent volume of distribution (V/F) - Period 2 | pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
  Pharmacokinetic variables

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided